CLINICAL TRIAL: NCT00005446
Title: Endogenous Estrogen and Coronary Heart Disease in Women
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4375; R29HL052123 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Postmenopausal women with coronary heart disease
- Postmenopausal women without coronary heart disease: Matched in age to the women with heart disease

SUMMARY:
To investigate the relation between endogenous levels of estrogen in postmenopausal women and the subsequent development of coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

Studies suggest that estrogen replacement therapy (ERT) lowers the risk of coronary heart disease in postmenopausal women. However, it is not known whether higher endogenous levels of estrogens in the postmenopausal period likewise have a protective effect.

DESIGN NARRATIVE:

The study used an existing resource of frozen blood samples from a cohort of 7,058 postmenopausal women enrolled between 1985 and 1991 for a study of endogenous hormones and cancer. The cohort was followed up to identify incident cases of coronary heart disease. One hundred thirty cases of coronary heart disease (defined as nonfatal myocardial infarction or death from coronary heart disease) were expected to occur by the end of follow-up. A nested case-control study was conducted in which each case was matched to two women from the cohort who were the same age as the case, donated blood around the same time, and were alive and free of heart disease as of the date of diagnosis of the case. Frozen serum samples from cases and their matched controls were analyzed for total estradiol, bioavailable estradiol (the estradiol fraction not bound to sex hormone binding globulin) estrone, total cholesterol, and high- and low-density lipoprotein cholesterol. Conditional logistic regression for matched sets were employed to determine whether estrogen levels were lower in the cases than their matched controls. The association between estrogen levels and cholesterol fractions was also investigated.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-04; Primary Completion 1999-03 (Actual)